CLINICAL TRIAL: NCT03002103
Title: An Open-label, Randomized, Controlled Phase III Trial Evaluating the Efficacy and Safety of EndoTAG®-1 in Combination With Paclitaxel and Gemcitabine Compared With Paclitaxel and Gemcitabine as First-line Therapy in Patients With Visceral Metastatic Triple-negative Breast Cancer
Brief Title: A Trial Evaluating the Efficacy and Safety of EndoTAG®-1 in Combination With Paclitaxel and Gemcitabine Compared With Paclitaxel and Gemcitabine as First-line Therapy in Patients With Visceral Metastatic Triple-negative Breast Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: study design reconsideration
Sponsor: SynCore Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT4005
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — MBT-0206; Paclitaxel; Gemcitabine

ARMS (2):
- ET+P+G (Experimental)
  Interventions: Drug: EndoTAG-1; Drug: Paclitaxel; Drug: Gemcitabine Hydrochloride
- Control (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: EndoTAG-1
  Arms: ET+P+G
Drug: Paclitaxel
Drug: Gemcitabine Hydrochloride

SUMMARY:
This is a prospective, multicenter, open-label, randomized, and controlled trial to test the superiority of EndoTAG®-1 in combination with paclitaxel and gemcitabine versus paclitaxel in combination with gemcitabine.

An independent data safety monitoring board (DSMB) will be established to decide on the recommended dose (RD) of EndoTAG®-1, paclitaxel and gemcitabine to be used throughout the trial and to monitor the patients' safety and treatment efficacy data

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Female
2. Age ≥ 18 years or legal age to provide informed consent according to local regulatory requirements.
3. Metastatic TNBC confirmed histologically by a certified local laboratory (or existing medical record for confirmation is acceptable for patients in the safety run-in stage) using archival paraffinated material from the original surgery specimens or from later materials, if available. Results of the certified local laboratory must be available to allow for randomization.

   Tumors should be considered negative for ER and PrR by immunohistochemistry (IHC) (< 1% positive tumor nuclei, as per American Society of Clinical Oncology/College of American Pathologists [ASCO/CAP] guideline recommendations, Hammond et al 2010) and negative for HER2 by IHC or fluorescent or chromogenic in situ hybridization (FISH or CISH). Patients with equivocal HER2 results by IHC should have the negativity status confirmed by FISH.
4. Patients must have had prior adjuvant treatment with either sequential or concurrent anthracycline- and/or taxane-based chemotherapy. Patients may have received neoadjuvant treatment prior to the adjuvant anthracycline- and/or taxane-based chemotherapy as well.

   Note: Neoadjuvant treatment alone is acceptable only for patients in the safety run-in stage.
5. Patients with a disease-free interval (DFI) on anthracycline- and/or taxane-based adjuvant therapy of ≥ 12 months.

   Note: This criteria is for main study only.
6. Patients must be indicated for treatment with polychemotherapy for visceral metastatic disease as judged by the Investigator.

   Note: Lymph node metastasis alone is acceptable only for patients in the safety run-in stage.
7. At least one measurable or non-measurable tumor lesion according to RECIST version 1.1 as assessed by the Investigator (local radiological image assessment).
8. ECOG performance status 0 or 1.
9. Negative pregnancy test (females of childbearing potential).
10. Willingness to perform double-barrier contraception during study and for 6 months post chemotherapy treatment (females of childbearing potential).
11. Signed informed consent.

Exclusion Criteria:

1. Prior first-line chemotherapy for locally recurrent and/or metastatic breast cancer, including visceral disease.
2. Brain metastasis/known progressive cerebral metastasis (patients with cerebral metastases in a stable state or after successful surgical or radiological treatment are allowed to participate in the study).
3. Major surgery < 4 weeks prior to enrollment.
4. Cancer immunotherapy at any time.
5. Severe pulmonary obstructive or restrictive disease.
6. Uncontrolled inflammatory disease (autoimmune or infectious).
7. Clinically significant cardiac disease (New York Heart Association [NYHA] stadium > 2).
8. Results of laboratory tests (hematology, coagulation, clinical chemistry) outside specified limits:

   * White blood cell (WBC) count ≤ 3 × 109/L
   * Absolute neutrophil count (ANC) ≤ 1.5 × 109/L
   * Platelets ≤ 100 × 109/L
   * Hemoglobin (Hb) ≤ 9.0 g/dL (≤ 5.6 mmol/L)
   * Activated partial thromboplastin time/international normalized ratio (aPTT/INR) > 1.5 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)> 2.5 × ULN (> 5 × ULN if presence of liver metastasis)
   * Alkaline phosphatase (AP) > 2 × ULN (> 5 × ULN if presence of liver metastasis)
   * Total bilirubin > 1.5 × ULN (> 2.5 × ULN if presence of liver metastasis)
9. Pregnancy or nursing status.
10. Known positive human immunodeficiency virus (HIV) infection in medical history.
11. Peripheral neuropathy associated to prior taxane therapy not recovered to grade 0 or 1.
12. Known hypersensitivity to any component of the EndoTAG®-1, standard paclitaxel and/or gemcitabine formulations.
13. History of malignancy other than breast cancer < 5 years prior to enrollment, except skin cancer (i.e., basal or squamous cell carcinoma) treated locally.
14. History of active or significant neurological disorder or psychiatric disorder that would prohibit the understanding and giving of informed consent, or would interfere in the clinical and radiological evaluation of central nervous system during the trial.
15. Concurrent treatment with other experimental products. Participation in another clinical trial with any investigational product within 30 days prior to study entry.
16. Positive test for hepatitis B (hepatitis B virus surface antigen [HBsAg] positive; or HBsAg negative but anti-hepatitis B virus core [HBc] antibody positive and HBV DNA positive) or hepatitis C (anti hepatitis C virus [HCV] antibody positive). Patients that are anti-HCV antibody positive can also be judged eligible if further HCV RNA detection shows negative results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2016-11-23 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 12 months
  Progression free survival defined as the time from randomization to disease progression based on blinded central radiological image evaluation according to response evaluation criteria in solid tumors (RECIST, version 1.1) or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall survival | 24 months
  from randomization to death from any cause
Clinical benefit rate | up to 24 months
Best overall tumor response rate | up to 24 months
  objective response or SD of any duration
Duration of response | up to 24 months
  the time from randomization to disease progression in the subgroup of patients responding to therapy
Quality of life(QLQ-C30,QLQ-BR23) | up to 24 months
  until disease progression
Post-progression PFS | up to 12 months
  as the time from start of second and subsequent lines of therapy administered after trial participation to disease progression (based on local radiological image evaluation or clinical assessment) or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Yi Chao, M.D., Ph.D., Principal Investigator — Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan
Locations (6):
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District